CLINICAL TRIAL: NCT06242327
Title: An Observational, Longitudinal Study to Describe the Outcome, and Outcome Predictors, of Patients With Primary Membranous Nephropathy, and the Nephrotic Syndrome Treated With Rituximab, or Other Monoclonal Antibodies
Brief Title: An Outcome Analysis of Primary Membranous Nephropathy
Acronym: PROMENADE
Status: Active, not recruiting | Type: Observational
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Other Study IDs: PROMENADE
Record Dates: First submitted 2024-01-25; First posted 2024-02-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Membranous Nephropathy
Keywords: Primary Membranous Nephropathy; Nephrotic Syndrome
MeSH Terms: conditions — Glomerulonephritis, Membranous; Nephrotic Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational study intended to track the course of the primary membranous nephropathy disease in real-world clinical practice.

The study will primarily assess the long-term outcomes of patients with primary membranous nephropathy in the context of advances in treatment options.

DETAILED DESCRIPTION:
Primary Membranous Nephropathy (PMN) is an autoimmune disease caused by the deposition of Immunoglobulin G and complement components on the subepithelial layer of the glomerular capillary wall. It affects 5-10 patients per million population and is the second cause of nephrotic syndrome in adults after diabetic kidney disease. For decades steroids and non-specific immunosuppressive medications have been advocated as a therapeutic option for patients with membranous nephropathy at increased risk of kidney failure because of persistent nephrotic syndrome. These medications, however, have major and potentially fatal adverse effects that offset their potential benefits and should be abandoned. Patients with PMN and non-nephrotic proteinuria (<3.5 g per 24 h) have a good prognosis with a supportive therapy based on optimized inhibition of the Renin-Angiotensin-System with Angiotensin-Converting-Enzyme inhibitors (ACEi) and/or Angiotensin-Receptor-Blockers (ARBs). Without immunosuppression, however, approximately one-third of patients with PMN and nephrotic syndrome (NS) (proteinuria >3.5 g per 24 h and/or hypoalbuminemia) progress to end stage kidney disease (ESKD). Steroids and non-specific immunosuppressive medications may achieve remission of the NS more effectively than placebo and supportive therapy but are associated with serious and potentially fatal complications that may offset the potential benefits of therapy. Thus, the 2012 Kidney Disease Improving Global Outcomes (KDIGO) guidelines recommended that the use of non- specific immunosuppressive therapy should be restricted to patients with persistent NS because, in this context, the reduced risk of ESKD could offset the risks of serious adverse events. The discovery of nephritogenic autoantibodies against podocyte M-type phospholipase A2 receptor (PLA2R) and thrombospondin type-1 domaincontaining protein 7A (THSD7A) antigens provided a clear pathophysiological rationale for interventions specifically targeting B cell lineages to prevent antibody production and subepithelial deposition. Anti-PLA2R antibody titer correlates with disease activity and patient outcome. Low autoantibody levels at diagnosis predict spontaneous remission, whereas high baseline anti-PLA2R antibody levels correlate with a reduced probability of spontaneous remission, are associated with progression to NS in patients with initial non-nephrotic proteinuria, and predict a high risk of relapse and progressive loss of kidney function. Moreover, decreasing anti-PLA2R antibody levels strongly predicts remission of proteinuria and response to various traditional and novel immunosuppressive treatments. Conceivably, in PLA2R-negative disease, PMN can be sustained by other nephritogenic autoantibodies such as anti-THSD7A antibodies that, similarly to anti-PLA2R antibodies, have been reported to predict disease activity and response to therapy.

Whether progression and response to treatment of patients with PMN can be affected not only by the overall titer of circulating anti-PLA2R autoantibodies, but also by their nature is matter of a lively debate. After almost 40 years of empirical treatment, the discovery of anti-PLA2R and anti-THSD7A autoantibodies provided the first clear pathophysiological rationale for interventions specifically aimed at preventing antibody production or their binding to specific antigens with subepithelial deposition of antibody-antigen immunocomplexes. The first-in-class anti-CD20 monoclonal antibody rituximab is safe and achieves remission in approximately two-thirds of patients with nephrotic membranous nephropathy. In PLA2R-related disease, remission is invariably preceded by depletion of anti PLA2R autoantibodies and relapse by their re-emergence into the circulation. Because of its superior risk/benefit profile as compared to non-specific immunosuppressive therapy, rituximab is now first-line therapy for patients with membranous nephropathy at risk of kidney failure. Novel monoclonal antibodies targeting CD20 cells (such as ofatumumab and obinutuzumab) and their differentiation (belimumab) or targeting long-living antibody producing CD38 memory cells (daratumumab, felzartamab) along with proteasome inhibitors such as bortezomib are being evaluated for the treatment of nephrotic patients with membranous nephropathy who are resistant or intolerant to rituximab. Complement inhibitor therapy might serve to stop the glomerular inflammatory process until the benefits of these medication become effective.

Researchers from the Department of Renal Medicine of Istituto di Ricerche Farmacologiche Mario Negri IRCCS, together with doctors from the Bergamo Hospital, were the first to document in 2002 that rituximab can recover totally or partially from the disease.

During the last twenty years, the Nephrology Unit of ASST-PG 23 (formerly, Ospedali Riuniti di Bergamo) become one of the most important disease specific Centers of excellence in the care of patients with PMN, more than 300 subjects were followed and treated with rituximab or other novel monoclonal antibodies in collaboration with "Centro di Ricerche Cliniche per le Malattie Rare Aldo e Cele Daccò", Ranica (BG) (Istituto Mario Negri IRCCS). The data collected at the routine visits of these patients represent an invaluable and unique source of information to describe the natural history of this rare disease and the evolution of the treatments. For this reason, we aim to create a data bank with the follow-up data of all the patients followed by the physicians of the Nephrology Unit in Bergamo and the Centro Daccò in Ranica who will agree to participate in the study and provide their consent to the use of their data for the research. Long-term data collection from a large patient sample may provide important insights regarding prognostic factors, characteristics of best responders to therapies, and estimation of the duration of unsuccessful treatment after which a patient can be considered a non-responder.

The variables evaluated in this study will complement and extend existing unknowledges on PMN, including provision of important information about the clinical course of the disease in patients receiving new treatments.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old) on the day of signing informed consent.
* Diagnosis of primary membranous nephropathy
* Nephrotic syndrome (proteinuria >3.5 g/24 hours)
* Written informed consent to the use of recorded data for research purposes.

Exclusion Criteria:

* Legal incapacity or limited legal capacity.
* Any contraindication to treatment with rituximab or other monoclonal antibody

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enrol all patients with a diagnosis of primary membranous nephropathy and the nephrotic syndrome (proteinuria >3.5 g/24-h) treated with rituximab or other monoclonal antibodies (including, among others, ofatumumab, obinutuzumab, felzartamab).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of disease remission | Through study completion, an average of 6 months
  Combined endpoint of complete (proteinuria < 0.3 g/24-hours) or partial (proteinuria <3 g/24-hours with >50% change vs proteinuria at baseline that is the time of the first rituximab or other monoclonal antibody administration) remission

SECONDARY OUTCOMES:
Evaluation of disease progression | Through study completion, an average of 6 months
  Assessment of disease progression and identification of the relevant disease outcome
Rate of GFR decline | Through study completion, an average of 6 months
  Rate of measured and estimated (CKD-Epi) GFR decline (or improvement)
Blood parameter levels | Through study completion, an average of 6 months
  Assessment of blood parameter levels considered as continuous variables
Incidence of adverse events | Through study completion, an average of 6 months
  Incidence of adverse events, as assessed and recorded in every-day clinical practice
Incidence of drug related adverse events | Through study completion, an average of 6 months
  Incidence of drug related adverse events, as assessed, and recorded in every-day clinical practice

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Remuzzi, MD, Study Director — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (2):
- Italy (2):
  - ASST HPG23 - Unità di Nefrologia, Bergamo, BG
  - Centro di Ricerche Cliniche per le Malattie Rare "Aldo e Cele Daccò", Ranica, BG

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schieppati A, Mosconi L, Perna A, Mecca G, Bertani T, Garattini S, Remuzzi G. Prognosis of untreated patients with idiopathic membranous nephropathy. N Engl J Med. 1993 Jul 8;329(2):85-9. doi: 10.1056/NEJM199307083290203. PMID 8510707
- [Background] Remuzzi G, Chiurchiu C, Abbate M, Brusegan V, Bontempelli M, Ruggenenti P. Rituximab for idiopathic membranous nephropathy. Lancet. 2002 Sep 21;360(9337):923-4. doi: 10.1016/S0140-6736(02)11042-7. PMID 12354476
- [Background] Ruggenenti P, Cravedi P, Chianca A, Perna A, Ruggiero B, Gaspari F, Rambaldi A, Marasa M, Remuzzi G. Rituximab in idiopathic membranous nephropathy. J Am Soc Nephrol. 2012 Aug;23(8):1416-25. doi: 10.1681/ASN.2012020181. Epub 2012 Jul 19. PMID 22822077
- [Background] Ruggenenti P, Debiec H, Ruggiero B, Chianca A, Pelle T, Gaspari F, Suardi F, Gagliardini E, Orisio S, Benigni A, Ronco P, Remuzzi G. Anti-Phospholipase A2 Receptor Antibody Titer Predicts Post-Rituximab Outcome of Membranous Nephropathy. J Am Soc Nephrol. 2015 Oct;26(10):2545-58. doi: 10.1681/ASN.2014070640. Epub 2015 Mar 24. PMID 25804280
- [Background] Ruggenenti P, Fervenza FC, Remuzzi G. Treatment of membranous nephropathy: time for a paradigm shift. Nat Rev Nephrol. 2017 Sep;13(9):563-579. doi: 10.1038/nrneph.2017.92. Epub 2017 Jul 3. PMID 28669992
- [Background] Perna A, Ruggiero B, Podesta MA, Perico L, Orisio S, Debiec H, Remuzzi G, Ruggenenti P. Sexual dimorphic response to rituximab treatment: A longitudinal observational study in a large cohort of patients with primary membranous nephropathy and persistent nephrotic syndrome. Front Pharmacol. 2022 Sep 2;13:958136. doi: 10.3389/fphar.2022.958136. eCollection 2022. PMID 36120314